CLINICAL TRIAL: NCT04902391
Title: A Multi-Disciplinary, Patient-Partnered, Pan-Canadian, Comparative Effectiveness Evaluation of an Innovative Acute Pediatric Mental Health and Addiction Care Bundle
Brief Title: A Patient-Partnered, Pan-Canadian, Comparative Effectiveness Evaluation of an Acute Pediatric Mental Health and Addiction Care Bundle
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: University of Alberta (Other); University of Saskatchewan (Other); University of Manitoba (Other); McMaster University (Other); Western University, Canada (Other); University of Toronto (Other); McGill University (Other); Dalhousie University (Other); Memorial University of Newfoundland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: REB20-1825
Record Dates: First submitted 2021-04-07; First posted 2021-05-26 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2024-12

CONDITIONS: Mental Health; Mental Disorders; Pediatrics; Emergency Psychiatric
Keywords: Emergency Psychiatric Services; Healthcare Delivery
MeSH Terms: conditions — Psychological Well-Being; Mental Disorders | interventions — Health Services

STUDY DESIGN:
Intervention Model Description: Pragmatic, parallel arm cluster randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acute Mental Health Care Bundle (Experimental): We developed an evidence-based bundle of care to address current gaps in care. The bundle: 1) brings together multiple evidence-based assessment tools (ASQ, HEADS-ED) to ensure efficient, high-value ED-based care; 2) removes barriers to assessment and builds connections to care: Assessments are conducted by a mental health care provider and families have access to urgent follow-up care; and 3) prioritizes family engagement: A shared decision-making framework (Choice and Partnership) is used to promote children and youth as stewards of their care and support partnership between EDs and follow-up services with the duration of care determined collaboratively by the patient and their provider.
  Interventions: Other: Health Services
- Usual ED-Based Mental Health Care (No Intervention): Local standards of ED-based mental health care will be delivered at control sites. Site leads have determined that this care does not involve the 3 specific core innovations in the bundle. Local care standards are similar across study sites and include use of CTAS score at triage (but no mental health risk assessment tool), ED physician medical clearance and assessment of consultation need, and no consistent mental health follow-up plan. Sites that are randomized to the control arm will not adopt core bundle elements.

INTERVENTIONS:
Other: Health Services — The Acute Mental Health Care Bundle consists of 3 core elements, including: (1) ED triage, (2) ED assessment and care, and (3) follow-up care.
  Arms: Acute Mental Health Care Bundle

SUMMARY:
The investigators will determine, in an 8-site, hybrid Type 1 cluster randomized effectiveness implementation trial, if an acute mental health care bundle, compared to standard care, improves wellbeing at 30 days in children and youth seeking emergency department care for mental health and substance use concerns.

DETAILED DESCRIPTION:
The investigators we co-designed, with parents and youth, an acute mental health care bundle-a set of evidence informed practices collectively used to improve the quality of care. The bundle of care includes:

1. Triage-based evaluation of risk for suicide [Ask Suicide-Screening Questions (ASQ) and HEADS-ED, an assessment mnemonic (Home; Education & Employment; Activities & Peers; Drugs & Alcohol; Suicidality; Emotions & Behaviours; Discharge or Current Resources]
2. Focused mental health team psychosocial evaluation to guide decision-making
3. Choice And Partnership Approach (CAPA) to care

This bundle of care also strives to remove the ED physician as the gatekeeper to mental health care and will facilitate, ideally, 24-48 hour urgent mental health follow-up (booked before the child/family leave the ED), with up to 96 hours to coordinate follow-up for patients attending the ED on weekends.

Primary Research Objective: To determine, in an 8-site, hybrid Type I cluster randomized effectiveness-implementation trial, if an acute mental health care bundle, compared to standard care, improves wellbeing at 30 days in children and youth seeking ED care for mental health and substance use concerns.

Secondary Research Objectives: (1) To determine if the bundle improves wellbeing, satisfaction with care, family functioning, and health care delivery; (2) To identify modifiable barriers, constraints, and enablers of bundle implementation fidelity and effectiveness; (3) To test if trial intervention effects are moderated by sociodemographic characteristics (sex, gender, ethnicity, culture, education, and socioeconomic status); and (4) To assess the cost-effectiveness of the approach.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8 to 17.99 years
2. Chief triage concern of at least one of the following (or comparable) mental health CEDIS triage categories:

   1. Anxiety/situational crisis and/or hyperventilation
   2. Bizarre/paranoid behaviour
   3. Concern for patient's welfare
   4. Depression/suicidal/deliberate self-harm
   5. Hallucinations/delusions
   6. Violent/homicidal behaviour
   7. Insomnia
   8. Pediatric disruptive behaviour

Exclusion Criteria:

1. Brought to the ED under provincial mental health legislation
2. Exhibiting features of schizophrenia, schizotypal, delusional disorders, or psychosis (e.g., hallucinations/delusions complaint should be reviewed carefully for this exclusion criterion)
3. Significant self-harm act (i.e., suicide attempt requiring medical clearance, excluding ideation or minor superficial wounds; e.g., laceration/puncture, overdose ingestion, etc.)
4. Other co-morbid medical concerns requiring oversight and/or medical clearance from an emergency physician (e.g., confusion/disorientation, substance withdrawal, other medical complaints, etc.)
5. Substance misuse/intoxication or altered level of consciousness
6. Exhibiting a behavioural syndrome associated with physiologic disturbances (e.g., anorexia)

   Children/youth will also be excluded based on language barriers:
7. Language barrier (i.e., patient and parent/legal guardian must be fluent in either English or French)

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6800 (Estimated)
Dates: Start 2022-02-09 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Warwick-Edinburgh Mental Wellbeing Scale 30 days after the index ED visit | 30 days after the index emergency department (ED) visit
  Measured in survey completed by the participant using the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) for patients ≥13 years
  Each item is scored on a range from 1 to 5. The total score will be between 14 and 70, with lower scores indicating poor wellbeing, and higher scores indicating greater wellbeing. Very low wellbeing is defined as a score of ≤ 45. A substantial decrease in wellbeing is a decrease by 5 or more points.
Stirling Children's Wellbeing Scale 30 days after the index ED visit | 30 days after the index emergency department (ED) visit
  Measured in survey completed by the participant using the Stirling Children's Wellbeing Scale (SCWBS) for patients <13 years.
  Each item is scored on a range from 1 to 5. The total score will be between 12 and 60, with lower scores indicating poor wellbeing, and higher scores indicating greater wellbeing. Very low wellbeing is defined as a score of ≤ 30. A substantial decrease in wellbeing is a decrease by 5 or more points.
  As these scales used for the primary outcomes measure the same construct, data will be standardized and combined across age groups to derive a single measure of wellbeing.

SECONDARY OUTCOMES:
Satisfaction with acute mental health care services as measured by the Service Satisfaction Scale 10 | 72 hours after the index ED visit
  Measured in survey completed by the participant using the Service Satisfaction Scale 10 (SSS-10). The scale consists of 12 items (parent version) or 10 items (youth version). Items are scored on a 5-point response scale with a total possible score of 60 (parent) or 50 (youth). Higher scores indicate higher satisfaction.
Quality of life as measured by the Beach Center Family Quality of Life Scale | 30 days after the index ED visit
  Measured in survey completed by the participant using the Beach Center Family Quality of Life Scale (FQOL). The 25-item scale uses a 5-point rating with a maximum score of 125 indicating highest quality of life.
Warwick-Edinburgh Mental Wellbeing Scale at 90 days after the index ED visit | 90 after the index ED visit
  Measured in survey completed by the participant using the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) for patients ≥13 years.
  Each item is scored on a range from 1 to 5. The total score will be between 14 and 70, with lower scores indicating poor wellbeing, and higher scores indicating greater wellbeing. Very low wellbeing is defined as a score of ≤ 45. A substantial decrease in wellbeing is a decrease by 5 or more points.
Stirling Children's Wellbeing Scale at 90 days after the index ED visit | 90 after the index ED visit
  Measured in survey completed by the participant using the Stirling Children's Wellbeing Scale (SCWBS) for patients <13 years.
  Each item is scored on a range from 1 to 5. The total score will be between 12 and 60, with lower scores indicating poor wellbeing, and higher scores indicating greater wellbeing. Very low wellbeing is defined as a score of ≤ 30. A substantial decrease in wellbeing is a decrease by 5 or more points.
  As the WEMWBS and SCWBS measure the same construct, data will be standardized and combined across age groups to derive a single measure of wellbeing.
Warwick-Edinburgh Mental Wellbeing Scale at 180 days after the index ED visit | 180 days after the index ED visit
  Measured in survey completed by the participant using the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) for patients ≥13 years.
  Each item is scored on a range from 1 to 5. The total score will be between 14 and 70, with lower scores indicating poor wellbeing, and higher scores indicating greater wellbeing. Very low wellbeing is defined as a score of ≤ 45. A substantial decrease in wellbeing is a decrease by 5 or more points.
Stirling Children's Wellbeing Scale at 180 days after the index ED visit | 180 days after the index ED visit
  Measured in survey completed by the participant using the Stirling Children's Wellbeing Scale (SCWBS) for patients <13 years.
  Each item is scored on a range from 1 to 5. The total score will be between 12 and 60, with lower scores indicating poor wellbeing, and higher scores indicating greater wellbeing. Very low wellbeing is defined as a score of ≤ 30. A substantial decrease in wellbeing is a decrease by 5 or more points.
  As the WEMWBS and SCWBS measure the same construct, data will be standardized and combined across age groups to derive a single measure of wellbeing.
Median duration of the index ED visits | Hours spent in the ED, measured at the index ED visit (Day 0)
  Measured using data collected in the patient electronic medical record. ED Length of stay is defined as the time interval between triage and discharge
Proportion of children and youth that revisited the emergency department for a mental health complaint related to their index emergency department visit within 7 and 30 days of the index visit | 7 and 30 days after the index ED visit
  Measured using data collected in the patient electronic medical record.
Proportion of emergency department visits for mental healthcare that concluded in hospital admission | Measured based on admissions following the index ED visit (Day 0)
  Measured using data collected in the patient electronic medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Freedman, MDCM, MSc, Principal Investigator — University of Calgary; Amanda Newton, PhD, Principal Investigator — University of Alberta
Locations (8):
- Canada (8):
  - The Children's Hospital of Winnipeg, Winnipeg, Manitoba
  - Janeway Children's Hospital, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - Jim Pattison Children's Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Derived] Rasiah J, Freedman S, Macdonald L, Prisnie K, Eltorki M, Finkelstein Y, Hopkin G, Santana MJ, Thull-Freedman J, Stang A, Prebeg M, Gagnon IJ, Steele M, Mater A, Katz L, Greenfield B, Plotnick L, Monga S, Lipman EL, Wright B, Dimitropoulos G, Porter R, Hurley K, Al Hamarneh YN, Newton A. Evaluation of parent and youth experiences in advisory groups as part of a mental healthcare clinical trial: protocol for a mixed-method study. BMJ Open. 2022 Jun 17;12(6):e059689. doi: 10.1136/bmjopen-2021-059689. PMID 35715176